CLINICAL TRIAL: NCT03593681
Title: The nCYT Study: A Powered Study to Evaluate the Sensitivity and Specificity of Cytological Evaluation of Fallopian Tube Samples Collected by the Cytuity in Determining the Presence of Malignancy
Brief Title: Compare Fallopian Tube Cells Collected by Cytuity With Removed Ovarian/Tubal Tissue to Determine Presence of Malignancy
Acronym: nCYT
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN 0507
Record Dates: First submitted 2018-07-10; First posted 2018-07-20 (Actual); Results first posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2020-12

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Ovarian Neoplasms; Ovary Cancer; Fallopian Tube Neoplasms; Fallopian Tube Adenocarcinoma; High Grade Serous Carcinoma; Peritoneal Carcinoma; Peritoneal Neoplasms; Adnexal Mass; Ovarian Diseases
Keywords: salpingo-oophorectomy; salpingectomy; ovarian cancer; fallopian tube cancer; high grade serous carcinoma; hysteroscopic biopsy; fallopian tube cell collection; peritoneal cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Peritoneal Neoplasms; Ovarian Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue and Cells
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Hysteroscopic cell sampling of the fallopian tube — Hysteroscopic fallopian tube biopsy
  Other Names: Cytuity

SUMMARY:
Prospective, multi-center, non-randomized study to assess the ability of the Cytuity device to collect cell samples from the fallopian tube that can be evaluated for the presence or absence of malignancy.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is medically cleared for surgery
2. Subject is scheduled to undergo salpingo-oophorectomy or salpingectomy for a pelvic mass suspicious for malignancy
3. Subject must be 18 years of age
4. Subject must be able to provide informed consent

Exclusion Criteria:

1. Contraindication to hysteroscopy
2. Acute pelvic inflammatory disease
3. Active or recent lower pelvic infection
4. Pregnancy
5. Delivery or termination of a pregnancy in the past 6 weeks
6. Known tubal obstruction
7. Tubal ligation
8. Invasive carcinoma of the cervix or endometrium
9. Intolerance of anesthesia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are scheduled to undergo a salpingo-oophorectomy or salpingectomy because of a pelvic mass suspicious for malignancy.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ted L Anderson, MD,PhD,FACOG, Principal Investigator — Vanderbilt University Medical Center
Locations (10):
- United States (10):
  - Scripps Clinic Medical Group, San Diego, California
  - Kaiser Permanente San Francisco Medical Center, San Francisco, California
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota
  - New York Presbyterian Hospital, New York, New York
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Scott & White Research Institute, Fort Worth, Texas
  - University of Virginia, Charlottesville, Virginia
  - Swedish Health Services, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Cytuity Cytological Evaluation: Those subjects enrolled in the study, with hysteroscope placed, ostia visualized, and adequate Cytuity cell sample collected.
Period: Overall Study
Arm/Group | Cytuity Cytological Evaluation
Started | 150
Completed | 115
Not Completed | 35
Not completed — Inadequate sample collected | 12
Not completed — Hysteroscope attempted but unable to find ostia | 11
Not completed — Protocol Violation | 3
Not completed — Withdrawal by Subject | 3
Not completed — Procedure not attempted | 3
Not completed — Adverse Event | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- Cytuity Cytological Evaluation: Subjects from whom a signed informed consent form was obtained.
Arm/Group | Cytuity Cytological Evaluation
Number analyzed (Participants) | 150
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age at Baseline | 53.9 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 3
  White | 125
  More than one race | 0
  Unknown or Not Reported | 10
Height [Mean (Standard Deviation); unit: cm] | 162.8 (7.9)
Weight [Mean (Standard Deviation); unit: kg] | 77.2 (21.3)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.1 (7.7)

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity and Specificity of Cytological Samples for Fallopian Tube Involvement
Description: Evaluate the sensitivity and specificity of the cytological samples collected from the fallopian tube in determining the presence or absence of malignancy for fallopian tube involvement as compared to the surgical histology results. Fallopian tube involvement was defined as: 1. Malignant cells that originated in the fallopian tube, detected by the surgical histology results from the fallopian tube. 2. Malignant cells that have migrated to the fallopian tube, detected by surgical histology results of the ovaries or fallopian tube.
Time Frame: At the time of the scheduled salpingectomy or salpingo-oophorectomy
Population: The number of Cytuity cell samples, not participants, was used for these endpoint analyses.
Measure: Number (95% Confidence Interval); unit: Proportion of Cytuity Cell Samples
Units Other Than Participants: Cytuity Cell Samples
Groups:
- Sensitivity - Proportion of Cytuity Cell Samples That Correctly Identify the Presence of Disease: The number of true positive Cytuity cell samples divided by the number of true positives and the number of false negatives.
- Specificity - Proportion of Cytuity Cell Samples That Correctly Identify the Absence of Disease: The number of true negative Cytuity cell samples divided by the number of true negatives and the number of false positives.
Arm/Group | Sensitivity - Proportion of Cytuity Cell Samples That Correctly Identify the Presence of Disease | Specificity - Proportion of Cytuity Cell Samples That Correctly Identify the Absence of Disease
Number analyzed (Participants) | NA | NA
Number analyzed (Cytuity Cell Samples) | 14 | 156
Proportion of Cytuity Cell Samples | .143 [.029 to .479] | .959 [.911 to .981]

2. Secondary Outcome: PPV, NPV and Diagnostic Accuracy for Fallopian Tube Involvement
Description: Positive Predictive Value, Negative Predictive Value and Diagnostic Accuracy will be calculated for Cytuity as compared to surgical histology of the ovaries and fallopian tube for fallopian tube involvement. Fallopian tube involvement was defined as: 1. Malignant cells that originated in the fallopian tube, detected by the surgical histology results from the fallopian tube. 2. Malignant cells that have migrated to the fallopian tube, detected by surgical histology results of the ovaries or fallopian tube.
Time Frame: At the time of the scheduled salpingectomy or salpingo-oophorectomy
Population: The number of Cytuity cell samples, not participants, was used for these endpoint analyses.
Measure: Number (95% Confidence Interval); unit: Proportion of Cytuity Cell Samples
Units Other Than Participants: Cytuity Cell Samples
Groups:
- PPV - Proportion of True Positive Results for Fallopian Tube Involvement: The proportion of positive Cytuity cell samples that came from a fallopian tube found to have histology positive for malignancy and/or a corresponding ovary found to have histology positive for malignancy
- NPV - Proportion of True Negative Results for Fallopian Tube Involvement: The proportion of negative Cytuity cell samples that came from a fallopian tube found to have histology negative for malignancy and a corresponding ovary found to have histology negative for malignancy
- Diagnostic Accuracy - Proportion of Accurate Diagnoses: The proportion of Cytuity cell sample results that conformed to the correct diagnosis as determined by the surgical histology results
Arm/Group | PPV - Proportion of True Positive Results for Fallopian Tube Involvement | NPV - Proportion of True Negative Results for Fallopian Tube Involvement | Diagnostic Accuracy - Proportion of Accurate Diagnoses
Number analyzed (Participants) | NA | NA | NA
Number analyzed (Cytuity Cell Samples) | 9 | 161 | 170
Proportion of Cytuity Cell Samples | 0.221 [0.032 to 0.71] | 0.932 [.877 to .963] | .894 [.834 to .934]

3. Secondary Outcome: Sensitivity, Specificity, PPV, NPV and Diagnostic Accuracy of the Fallopian Tube
Description: Sensitivity, Specificity, Positive Predictive Value, Negative Predictive Value and Diagnostic Accuracy will be calculated for Cytuity as compared to surgical histology of the fallopian tube.
Time Frame: At the time of the scheduled salpingectomy or salpingo-oophorectomy
Population: The number of Cytuity cell samples, not participants, was used for these endpoint analyses.
Measure: Number (95% Confidence Interval); unit: Proportion of Cytuity Cell Samples
Units Other Than Participants: Cytuity Cell Samples
Groups:
- Sensitivity - Proportion of Cytuity Cell Samples That Correctly Identify the Presence of Disease: The number of true positive Cytuity cell samples divided by the number of true positive and the number of false negatives
- PPV - Proportion of True Positive Results for Fallopian Tube Pathology: The proportion of positive Cytuity cell samples that came from a fallopian tube also found to have histology positive for malignancy
- NPV - Proportion of True Negative Results for Fallopian Tube Pathology: The proportion of negative Cytuity cell samples that came from a fallopian tube also found to have histology negative for malignancy
Arm/Group | Sensitivity - Proportion of Cytuity Cell Samples That Correctly Identify the Presence of Disease | Specificity - Proportion of Cytuity Cell Samples That Correctly Identify the Absence of Disease | PPV - Proportion of True Positive Results for Fallopian Tube Pathology | NPV - Proportion of True Negative Results for Fallopian Tube Pathology | Diagnostic Accuracy - Proportion of Accurate Diagnoses
Number analyzed (Participants) | NA | NA | NA | NA | NA
Number analyzed (Cytuity Cell Samples) | 13 | 157 | 9 | 161 | 170
Proportion of Cytuity Cell Samples | .077 [.008 to .467] | .952 [.903 to .977] | .108 [.008 to .652] | .932 [.877 to .963] | .888 [.826 to .929]

4. Secondary Outcome: Sensitivity, Specificity, PPV, NPV and Diagnostic Accuracy of the Ovaries
Description: Sensitivity, Specificity, Positive Predictive Value, Negative Predictive Value and Diagnostic Accuracy will be calculated for Cytuity as compared to surgical histology of the ovaries for epithelial malignancies.
Time Frame: At the time of the scheduled salpingectomy or salpingo-oophorectomy
Population: The number of Cytuity cell samples, not participants, was used for these endpoint analyses.
Measure: Number (95% Confidence Interval); unit: Proportion of Cytuity Cell Samples
Units Other Than Participants: Cytuity Cell Samples
Groups:
- Sensitivity - Proportion of Cytuity Cell Samples That Correctly Identify the Presence of Disease: Number of true positive Cytuity cell samples divided by the number of true positives and the number of false negatives
- PPV - Proportion of True Positive Results for Ovary Pathology for Epithelial Malignancy: The proportion of positive Cytuity cell samples that came from a fallopian tube adjacent to a corresponding ovary found to have histology positive for malignancy
- NPV - Proportion of True Negatives for Ovary Pathology for Epithelial Malignancy: The proportion of negative Cytuity cell samples that came from a fallopian tube adjacent to a corresponding ovary found to have histology truly negative for malignancy
Arm/Group | Sensitivity - Proportion of Cytuity Cell Samples That Correctly Identify the Presence of Disease | Specificity - Proportion of Cytuity Cell Samples That Correctly Identify the Absence of Disease | PPV - Proportion of True Positive Results for Ovary Pathology for Epithelial Malignancy | NPV - Proportion of True Negatives for Ovary Pathology for Epithelial Malignancy | Diagnostic Accuracy - Proportion of Accurate Diagnoses
Number analyzed (Participants) | NA | NA | NA | NA | NA
Number analyzed (Cytuity Cell Samples) | 22 | 135 | 7 | 150 | 157
Proportion of Cytuity Cell Samples | .091 [.02 to .331] | .963 [.913 to .985] | .281 [.04 to .788] | .883 [.812 to .929] | .851 [.779 to .902]

5. Secondary Outcome: Sensitivity, Specificity, PPV, NPV and Diagnostic Accuracy for Subject Level Analysis
Description: Sensitivity, Specificity, Positive Predictive Value, Negative Predictive Value and Diagnostic Accuracy will be calculated for Cytuity as compared to surgical histology for fallopian tube involvement at the subject level. Fallopian tube involvement was defined as: 1. Malignant cells that originated in the fallopian tube, detected by the surgical histology results from the fallopian tube. 2. Malignant cells that have migrated to the fallopian tube, detected by surgical histology results of the ovaries or fallopian tube.
Time Frame: At the time of the scheduled salpingectomy or salpingo-oophorectomy
Measure: Count of Participants; unit: Participants
Groups:
- Sensitivity - Subjects in Which the Cytuity Correctly Identified the Presence of Disease: Number of subjects with true positive Cytuity cell samples divided by the number of subjects with true positives and the number of subjects with false negatives
- Specificity - Subjects in Which the Cytuity Correctly Identified the Absence of Disease: The number of subjects with true negative Cytuity cell samples divided by the number of subjects with true negatives and the number of subjects with false positives
- PPV - True Positive Results for Fallopian Tube Involvement on Subject Level: The number of subjects with a positive Cytuity cell sample and a fallopian tube and/or corresponding ovary with histology positive for malignancy
- NPV - True Negative Results for Fallopian Tube Involvement on Subject Level: The number of subjects with a negative Cytuity cell sample and a fallopian tube and corresponding ovary with histology negative for malignancy
- Diagnostic Accuracy - Subjects With Accurate Diagnoses: The number of subjects with a Cytuity cell sample result that conformed to the correct diagnosis on a subject level as determined by the surgical histology results
Arm/Group | Sensitivity - Subjects in Which the Cytuity Correctly Identified the Presence of Disease | Specificity - Subjects in Which the Cytuity Correctly Identified the Absence of Disease | PPV - True Positive Results for Fallopian Tube Involvement on Subject Level | NPV - True Negative Results for Fallopian Tube Involvement on Subject Level | Diagnostic Accuracy - Subjects With Accurate Diagnoses
Number analyzed (Participants) | 10 | 64 | 8 | 66 | 74
Participants | 2 | 58 | 2 | 58 | 60

ADVERSE EVENTS:
Time Frame: Adverse events occurring from the time the hysteroscope entered the subject until study exit (defined as 24 hours post-Cytuity use or discharge, whichever occurs first).
Groups:
- Treated Subjects: Subjects who signed the informed consent and had hysteroscope placement attempted
Arm/Group | Treated Subjects
All-Cause Mortality (participants affected / at risk) | 0/130
Serious Adverse Events (participants affected / at risk) | 3/130
Other Adverse Events (participants affected / at risk) | 2/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treated Subjects (N=130)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treated Subjects (N=130)
Uterine Perforation (Injury, poisoning and procedural complications) | 1 (1)
Fallopian Tube perforation (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-22): https://cdn.clinicaltrials.gov/large-docs/81/NCT03593681/Prot_SAP_000.pdf